CLINICAL TRIAL: NCT06394830
Title: A Phase 2b, Open Label, Single-Arm, Multi-Center, Multiple Dose, 14-Day Study to Evaluate the Safety, Efficacy, and Frequency of Intravesical Administration of VNX001 in Acute Treatment of Subjects With Interstitial Cystitis/Bladder Pain Syndrome (IC/BPS) Who Have an Episode of Acute Bladder Pain of Moderate to Severe Intensity
Brief Title: Safety, Efficacy, and Frequency of Administration of VNX001 in the Treatment of Interstitial Cystitis / Bladder Pain Syndrome (IC/BPS)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Vaneltix Pharma, Inc. (Industry)
Collaborators: Prevail Infoworks (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VNX001-110
Record Dates: First submitted 2024-04-24; First posted 2024-05-01 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Interstitial Cystitis; Bladder Pain Syndrome
Keywords: interstitial cystitis (IC); bladder pain syndrome (BPS); alkalinized lidocaine; heparin; intravesical; VNX001
MeSH Terms: conditions — Cystitis, Interstitial

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Open Label Arm (Experimental): VNX001 intravesical administration PRN up to 6 doses over 14 days. The VNX001 effective dose is 15 mL of buffered lidocaine HCl (200 mg) and sodium heparin (50,000 USPU).
  Interventions: Drug: VNX001

INTERVENTIONS:
Drug: VNX001 — Intravesical administration of VNX001

SUMMARY:
This is an open-label study that will enroll participants with Interstitial Cystitis / Bladder Pain Syndrome (IC/BPS).

The study will assess PRN (as needed) dosing of up to 6 intravesical (via catheter) doses of VNX001 (study drug) to treat acute instances of moderate to severe bladder pain over a 14-day period. The main aim of the study is to tally the number of doses and assess pain before and after doses. The study will review the safety and tolerability of VNX001.

Participants will need to attend up to seven (7) clinic visits (1 for screening and up to 6 visits for VNX001 dosing) or at least one (1) clinic visit (for a combined screening/dosing visit) and 5 telephone visits over the course of 14 days. Participants will also be asked complete a diary or telephone call each day of the study, in order to record bladder pain, urinary urgency, side effects, and medications taken.

ELIGIBILITY:
Inclusion Criteria:

1. Enrolled and completed Study VNX001-111 (i.e., at any site that is concurrently conducting the VNX001-111 study, a subject must have previously enrolled and completed Study VNX001-111 to be eligible for entry into the VNX001-110 study) and meet all other inclusion/exclusion criteria.
2. Be able and willing to give a signed informed consent and to follow study instructions.
3. Be male or female, ≥ 18 years of age.
4. Have a history of IC/BPS for at least 9 months prior to the study, either treated (e.g. Elmiron®, RIMSO-50®), or untreated.
5. Have received a cystoscopy in association with their diagnosis of IC/BPS within 1 year of screening.
6. Have a score of ≥ 14 and ≤ 30 on the PUF questionnaire, completed at screening.
7. Have an episode of acute bladder pain of moderate to severe intensity with a minimum score of 4 on the 11-point bladder pain NRS at time of screening and 15 minutes post void immediately prior to study drug administration.

Exclusion Criteria:

1. For females, have a positive pregnancy test at screening or be pregnant or lactating.

   Note: Females considered to be of child-bearing potential must commit to using a consistent and medically acceptable method of birth control for the duration of the study: hormonal (i.e., oral, transdermal patch, implant, or injection) on a stable dose for at least 3 months prior to screening; double barrier (i.e., condom with spermicide or diaphragm with spermicide) consistently for at least 2 weeks prior to screening; and intrauterine device for at least 3 months prior to screening; or only have a partner who has been vasectomized for at least 6 months prior to screening or exclusively has same-sex partners. Female participants who are abstinent from heterosexual intercourse as part of their usual lifestyle will also be eligible for participation. Females considered to be of non-childbearing potential include: At least 1 year postmenopausal; surgically sterile (tubal ligation, bilateral oophorectomy, salpingectomy, of hysterectomy); congenitally sterile; diagnosed as infertile and not undergoing treatment to reverse infertility.
2. Males who are sexually active with females and are not willing to commit to an acceptable method of birth control for the duration of the study.
3. Postmenopausal women who, if taking hormone replacement therapy, have not been stabilized on a regimen of hormone replacement therapy within 3 months of screening.
4. Have a known hypersensitivity to heparin or lidocaine.
5. Have used any local anesthetic by any route (other than intravesical instillation) within 48-hours prior to study drug administration, or used a lidocaine patch or lidocaine containing topical compounds within 14 days prior to study drug administration.
6. Have used a tricyclic antidepressant, or a gamma-aminobutyric acid (GABA) analogue (gabapentin or pregabalin), unless taking a stable dose of the medication for ≥ 3 weeks. The stable dose of gabapentin may not exceed 1,200 mg per day, and the stable dose of pregabalin may not exceed 150 mg per day.
7. Have used prohibited drugs as determined by self-report, positive urine drug screen, or in the opinion of the investigator be under the influence of drugs affecting mentation precluding their ability to follow the study protocol or bias study results.
8. Have a known abnormal laboratory test value that, in the investigator's judgement, is clinically significant.
9. Have a neurogenic bladder or other disorder that, in the opinion of the investigator, may cause neurogenic bladder (including Parkinson's disease, multiple sclerosis, epilepsy, myasthenia gravis, movement disorders, spinal cord damage).
10. Have pain or a pain disorder that, in the opinion of the investigator, would make it difficult to discriminate pelvic pain of bladder origin from the other pain.
11. Have any of the following central nervous system (CNS) conditions that in the opinion of the investigator would impact the subject's study participation due to their ability to follow the study protocol or bias study results, severe diagnosed: major depressive disorder, bipolar disorder, schizophrenia, general anxiety disorder, attention deficit disorder, obsessive compulsive disorder, or other major CNS disorder.
12. Have history of arrhythmias, conduction disturbances, or cardiac disease, or any coexisting medical condition that, in the opinion of the investigator, may be significant or interfere with study procedures or interpretation of study results.
13. Had bladder instillation therapy within 14 days prior to study entry.
14. Had an in-office cystoscopy within 7 days prior to study drug administration.
15. Had dilatation (hydrodistension) of bladder within 3 months of study entry.
16. Evidence or suspected presence of cancer detected during cystoscopy.
17. Has received any investigational drug or device within 30 days prior to screening.
18. Is currently enrolled in another investigational drug or device study.
19. Is unwilling or unable to abide by the requirements of the study.
20. Have an actively bleeding lesion or area in the bladder as detected by dipstick urinalysis and investigator assessment, immediately prior to randomization (Section 9.5.1.6). If the investigator determines that active bleeding is not occurring and that it is safe for the subject, the subject may continue in the study.
21. Have a history of coagulopathy or taking anticoagulants.
22. Are taking any of the following medications:

    * Phenytoin
    * Carbamazepine
    * St. John's Wort
    * Phenobarbital
    * Rifampin
23. Have had any of the following:

    * Bacterial cystitis within 30 days as demonstrated by a positive urine culture (≥ 105 bacteria per mL)
    * History of pelvic irradiation or radiation cystitis
    * History or presence of uterine, cervical, pelvic, rectal, ovarian, or vaginal cancer
    * History of benign or malignant bladder tumors
    * Current chemotherapy
    * History or presence of tuberculous cystitis
    * History or presence of chemical cystitis, including that due to cyclophosphamide
    * History or presence of urinary schistosomiasis
    * Bladder or ureteral calculi
    * Clinically significant infectious vaginitis
    * Currently uncontrolled genital herpes
    * History or presence of urethral diverticulum
    * Presence of bladder fistulae
    * History of ketamine use

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-12-13 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Frequency of PRN intravesical administrations of VNX001 | 14 Days

SECONDARY OUTCOMES:
Change in bladder pain from first dose baseline to 1, 2, 6, 12, and 24 hours post-dose | Through 24 Hours
  Average absolute change and average percentage change in bladder pain from baseline to 1, 2, 6, 12, and 24 hours post-dose, as determined using an 11-point numerical rating scale (NRS) for bladder pain. The 11-point NRS for bladder pain is a scale from 0 to 10, with 0 indicating no bladder pain and 10 indicating the worst imaginable bladder pain.
Change in bladder pain after each repeat dose to 1, 6, 12, and 24 hours post-dose | Through 24 Hours
  Average absolute change and average percentage change in bladder pain from after each repeat dose to 1, 6, 12, and 24 hours post-dose, as determined using an 11-point numerical rating scale (NRS) for bladder pain. The 11-point NRS for bladder pain is a scale from 0 to 10, with 0 indicating no bladder pain and 10 indicating the worst imaginable bladder pain.
Sum of bladder pain intensity differences from baseline to 6, 10, and 24 hours post-dose (SPID-6, SPID-10, and SPID-24, respectively) | Through 24 Hours
  A measure of the sum of bladder pain intensity differences from baseline to 6, 10, and 24 hours post-dose (SPID-6, SPID-10, and SPID-24, respectively), as determined using an 11-point numerical rating scale (NRS) for bladder pain. The 11-point NRS for bladder pain is a scale from 0 to 10, with 0 indicating no bladder pain and 10 indicating the worst imaginable bladder pain.
Change in the Patient Overall Rating of Improvement of Symptoms (PORIS) questionnaire | Through 24 Hours
  Change in percentage of subjects achieving ≥ 50% improvement in pain, urgency and overall improvement using the PORIS questionnaire at 1, 12, and 24 hours post-dose. The PORIS questionnaire is an assessment of the subject's condition after treatment compared to before treatment. Subjects will be asked to select the category that best describes the overall change in their condition compared to before receiving study medication; the choices are: worse, no better (0% improvement), slightly improved (25% improvement), moderately improved (50% improvement), greatly improved (75% improvement), or symptoms gone (100% improvement).
Pain scale threshold associated with subjects seeking repeat dosing | 14 Days
  The average NRS pain assessment threshold before each PRN repeat intravesical VNX001 treatment. The 11-point NRS for bladder pain is a scale from 0 to 10, with 0 indicating no bladder pain and 10 indicating the worst imaginable bladder pain.
Adverse events (AEs) | up to 17 Days
  Incidence of treatment-emergent adverse events (TEAEs), drug-related adverse events (AEs), and discontinuations due to AEs through the last follow up call at 48-72 hours after the last clinic or telephone visit.

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Arizona Urology Specialists, Tucson, Arizona
  - Valley Urology, Inc., Fresno, California
  - Prestige Medical Group, Tustin, California
  - Georgia Urology, Cartersville, Georgia
  - Oregon Urology Institute, Springfield, Oregon

IPD SHARING:
Plan to Share IPD: No